CLINICAL TRIAL: NCT02574351
Title: Study of T-Regulatory Cells in Asthma
Status: Completed | Type: Observational
Sponsor: Northwell Health (Other)
Responsible Party: Sponsor
Other Study IDs: 11-076B
Record Dates: First submitted 2013-11-01; First posted 2015-10-12 (Estimated); Last update posted 2016-01-29 (Estimated); Status verified 2016-01

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — Blood Specimen Collection

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — T regulatory cells are isolated in the blood specimens
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- obese asthmatic: Participants from this group will be included in this study. A blood draw, breathing test will be performed to see if there is a difference in the t-regulatory cells amongst this group.
  Interventions: Biological: blood draw, breathing test
- normal asthmatic: Participants from this group will be included in this study. A blood draw, breathing test will be performed to see if there is a difference in the t-regulatory cells amongst this group
  Interventions: Biological: blood draw, breathing test
- obese control: Participants from this group will be included in this study. A blood draw, breathing test will be performed to see if there is a difference in the t-regulatory cells amongst this group.
  Interventions: Biological: blood draw, breathing test
- normal control: Participants from this group will be included in this study. A blood draw, breathing test will be performed to see if there is a difference in the t-regulatory cells amongst this group.
  Interventions: Biological: blood draw, breathing test

INTERVENTIONS:
Biological: blood draw, breathing test — A blood draw,breathing test will be performed on every participant

SUMMARY:
To study whether the immune response as directed by regulatory T cells is different between obese asthmatics, normal weight asthmatics and healthy controls.

DETAILED DESCRIPTION:
The investigators hypothesize that the increase in asthma severity in obese patients is, at least in part, related to a defective number or function of regulatory T cells (Tregs). That is in the obese asthmatic subject a defective Treg profile would augment the inflammation of asthma (a synergistic effect). Alternatively, that Treg dysfunction in obesity might affect asthma independently (an additive effect). To test these hypotheses, the investigators plan to conduct an observational controlled study to compare Treg profile in obese and normal-weight individuals with and without asthma.

This is an exploratory study to investigate the following:

1. To determine whether Treg number and function differs between obese and normal-weight individuals with and without asthma.
2. To determine whether serum leptin levels differ between obese and normal-weight individuals with and without asthma.

ELIGIBILITY:
Inclusion Criteria:

1. Obese asthmatics
2. Normal weight asthmatics
3. Healthy obese
4. Health non-obese

Asthmatic subjects will be recruited:

1. If they have a physician diagnosis of adult onset asthma (asthma diagnosed after the age of 18).
2. If they have stable disease without exacerbation, physician or emergency department visits, or change in asthma medication for the past 4 weeks, inhaled steroids will be allowed.

Non asthmatic subjects

1. Will not have had a prior diagnosis of asthma,
2. Have no history of atopy.
3. Have no history of lung diseases.

Exclusion Criteria:

1. > 10 pack year smoking history, or currently smoking
2. Pulmonary disease other than asthma.
3. History of heart disease
4. Weight loss greater than 10 kg, or greater than 10% initial body weight within the past 3 months.
5. Any agents that could potentially alter the inﬂammatory system such as thiazolidinedione, a statin, or oral steroid therapy.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Females in good health between the ages of 18-50, with or without asthma.
Sampling Method: Non-Probability Sample
Enrollment: 66 (Actual)
Dates: Start 2011-05; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Difference of treg and serum leptin levels among obese and normal weight individuals with and without asthma. | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Rubin Cohen, MD, Principal Investigator — North Shore
Locations (1):
- North Shore LIJ Health System, New Hyde Park, New York, United States